CLINICAL TRIAL: NCT02137590
Title: An Open Label Pilot Study to Evaluate the Efficacy of Spanish Black Radish on the Induction of Phase I and Phase II Enzymes in Healthy Male Subjects
Brief Title: An Open Label Pilot Study to Evaluate the Efficacy of Spanish Black Radish on the Induction of Phase I and Phase II Enzymes
Acronym: 11SEHS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11SEHS
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Spanish Black Radish; Phase I detoxification enzymes; Phase II detoxification enzymes; Acetaminophen

ARMS (1):
- Spanish Black Radish (Experimental): Spanish Black Radish product
  Interventions: Dietary Supplement: Spanish Black Radish product

INTERVENTIONS:
Dietary Supplement: Spanish Black Radish product

SUMMARY:
This study will investigate the effect of Spanish Black Radish on phase I and phase II enzyme activity in healthy adult males. The primary objective is to determine the effect on phase I and phase II enzyme activity by measuring plasma and urine acetaminophen metabolite concentrations prior to and after a 28 day supplementation period with Spanish black radish product.

ELIGIBILITY:
Inclusion Criteria:

* Male age 25 - 35 years
* BMI 18 - 25 kg/m2
* Healthy as determined by laboratory results, medical history
* Agrees to avoid the consumption of cruciferous vegetables for 14 days prior to baseline and during the study treatment period
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Chronic diseases or any medical conditions
* Gall bladder disorders and /or bowel obstruction
* Use of prescribed or over the counter medications for the treatment of any acute or chronic conditions
* Use of muscle building steroids or body building aids
* Use of products containing ingredients derived from the Cruciferae (Brassicaracea) plant family within 14 days prior to randomization
* Use of natural health products other than vitamins or minerals within 14 days prior to randomization
* Any clinically significant abnormal laboratory value. Meaning a disease process, an exacerbation or worsening of an existing condition, requires further or more frequent monitoring or requires further action(s) to be taken. Clinical significance can only be determined by the Qualified Investigator.
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to test product ingredients, Cruciferae/Brassicaracea plant family (includes mustard, cabbage, radish), acetaminophen or foods and beverages provided during the study
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
* Cannot take acetaminophen within 48 hrs of the baseline appointment or final 4-wk appointment.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect on Phase I and II enzymes | 4 weeks
  The effect on phase I and phase II enzyme activity determined by measuring plasma and urine acetaminophen metabolite concentrations Subjects will ingest 1000 mg of acetaminophen. Blood will be collected at 0, 2, 4, 6 and 8 hours after acetaminophen dosage for the analysis of plasma acetaminophen metabolites. These measurements will be performed prior to and after 4 weeks of treatment with Spanish Black Radish product.

SECONDARY OUTCOMES:
Assessment of Hormone Levels | 4 weeks
  Assessment of serum total testosterone, free testosterone and estradiol 17 beta

OTHER OUTCOMES:
Blood Safety Parameters | 4 weeks
  Assessment of CBC, electrolytes (Na, K, Cl), creatinine, AST, ALT, GGT, and bilirubin
Vital Signs | 4 weeks
  Assessment of Blood Pressure and Heart Rate
Adverse Events | 4 weeks
  Assessment of any adverse events occurring during the study

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.; Malkanthi Evans, PhD, Study Director — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada

REFERENCES:
- [Derived] Evans M, Paterson E, Barnes DM. An open label pilot study to evaluate the efficacy of Spanish black radish on the induction of phase I and phase II enzymes in healthy male subjects. BMC Complement Altern Med. 2014 Dec 9;14:475. doi: 10.1186/1472-6882-14-475. PMID 25490898